CLINICAL TRIAL: NCT04909489
Title: Study on the Characteristics of Phlegm-Dampness Retention Syndrome and the Spleen and Kidney Yang Deficiency of Dyslipidemia From the Oxidative Stress Enhancement Caused by Inhibition of Serine Metabolic Pathway
Brief Title: PDR and SKYD of Dyslipidemia's Characteristics From the Oxidative Stress Enhancement Caused by Inhibition of Serine Metabolic Pathway
Acronym: PDR SKYD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dongzhimen Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Chao Ye, Principal Investigator, Dongzhimen Hospital, Beijing
Other Study IDs: 2021DZMEC-047-02
Record Dates: First submitted 2021-05-23; First posted 2021-06-01 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Traditional Chinese Medicine; Dyslipidemias; Syndrome
Keywords: metabonomics; syndrome; dislipidemia; serine metabolic pathway; Chinese medicine; PHGDH
MeSH Terms: conditions — Dyslipidemias; Syndrome | interventions — Cross-Sectional Studies; Methods

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PDR group: Phlegm-Dampness Retention syndrome group
  Interventions: Other: cross-sectional study without intervention
- SKYD group: Spleen and Kidney Yang Deficiency syndrome group
  Interventions: Other: cross-sectional study without intervention
- NC group: Normal Control group
  Interventions: Other: cross-sectional study without intervention

INTERVENTIONS:
Other: cross-sectional study without intervention — cross-sectional study without intervention

SUMMARY:
Clinical epidemiological investigation and modern statistics will be used. Syndrome was quantified by TCM syndrome score scale. Metabonomics, proteomics, transcriptomics, enzyme-linked immunosorbent assay, xanthine oxidation method and thiobarbital method will be used to detect the relevant indicators in serum, urine and tongue coating, and "disease syndrome cell model" will be constructed to detect the relevant indicators. Objective to clarify the epigenetic basis, molecular biological regulation mechanism and core function characteristics of phgdh expression decline caused by PDR and SKYD of dyslipidemia, analyze the correlation between phgdh, serine metabolic pathway product concentration and oxidative stress level, and reveal the scientific connotation of the disease syndrome.

DETAILED DESCRIPTION:
Clinical epidemiological investigation and modern statistics will be used. Syndrome was quantified by TCM syndrome score scale. Metabonomics, proteomics, transcriptomics, enzyme-linked immunosorbent assay, xanthine oxidation method and thiobarbital method will be used to detect the relevant indicators in serum, urine and tongue coating, and "disease syndrome cell model" will be constructed to detect the relevant indicators. Objective to clarify the epigenetic basis, molecular biological regulation mechanism and core function characteristics of phgdh expression decline caused by PDR and SKYD of dyslipidemia, analyze the correlation between phgdh, serine metabolic pathway product concentration and oxidative stress level, and reveal the scientific connotation of the disease syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. inclusion criteria of dyslipidemia with SKYD and PDR. (1) subjects with dyslipidemia in accordance with the diagnostic standards and TCM syndrome diagnostic standards, (2) ranged in age from 20 to 80, (3) who signed the informed consent, and (4) without lipid-lowering medications.
2. inclusion criteria of NC. (1) healthy subjects, (2) ranged in age from 20 to 80, (3) who signed the informed consent.

Exclusion criteria:

Exclusion criteria of dyslipidemia with SKYD and PDR. The exclusion criteria were composed of four criteria and a patient was excluded if they fails on any of the criteria. Mentioned criteria were: (1) secondary dyslipidemia (causes of dyslipidemia include but not limited to hypothyroidism, nephrotic syndrome, chronic renal failure, liver diseases, diseases of the hematopoietic system, adrenal-corticosteroid or contraceptive-drug induced dyslipidemia); (2) aphasias, and patients had difficulties to speak or unable to extend tongue for tongue observation; (3) patients with psychosis or unable to answer questions properly; (4) patients with acute infectious diseases or in the acute disease states (such as acute myocardial infarction, acute cerebrovascular disease, etc.), as well as pregnant women.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In this study, 240 patients meet the inclusion criteria, including 100 cases of SKYD group and 100 cases of PDR group. Another 40 cases are NC group.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2021-04-21 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Routine Blood Examination | 2 years
  PDR group, SKYD group and NC group's Routine Blood Examination
Blood Biochemistry | 2 years
  PDR group, SKYD group and NC group's Blood Biochemistry
Routine Urine Examination | 2 years
  PDR group, SKYD group and NC group's Routine Urine Examination
the Methylation Level of PHGDH | 2 years
  Methylation sensitive restriction enzyme technique combined with PCR (msre-pcr) will be used to detect the Methylation Level of PHGDH in PDR group, SKYD group and NC group.
the Methylation Level of PHGDH in the cell models of disease-TCM syndrome | 2 years
  Methylation sensitive restriction enzyme technique combined with PCR (msre-pcr) will be used to detect the Methylation Level of PHGDH in the cell models of disease-TCM syndrome.
Distribution of h3k4me3, H3K9Ac and h3k27ac histones in PHGDH gene promoter | 2 years
  The distribution of h3k4me3, H3K9Ac and h3k27ac histones in the promoter of PHGDH gene will be detected by chromatin immunoprecipitation assay (chip) in PDR group, SKYD group and NC group.
Distribution of h3k4me3, H3K9Ac and h3k27ac histones in PHGDH gene promoter in the cell models of disease-TCM syndrome | 2 years
  The distribution of h3k4me3, H3K9Ac and h3k27ac histones in the promoter of PHGDH gene will be detected by chromatin immunoprecipitation assay (chip) in the cell models of disease-TCM syndrome.
3-phosphoglycerate dehydrogenase (PHGDH) RNA | 2 years
  PHGDH RNA level will be detected by fluorescence quantitative PCR in PDR group, SKYD group and NC group.
3-phosphoglycerate dehydrogenase (PHGDH) RNA in the cell models of disease-TCM syndrome | 2 years
  PHGDH RNA level will be detected by fluorescence quantitative PCR in the cell models of disease-TCM syndrome.
Phosphoserine aminotransferase (PSAT1) RNA | 2 years
  PSAT1 RNA level will be detected by fluorescence quantitative PCR in the cell models of disease-TCM syndrome.
Phosphoserine aminotransferase (PSAT1) RNA in the cell models of disease-TCM syndrome | 2 years
  PSAT1 RNA level will be detected by fluorescence quantitative PCR in the cell models of disease-TCM syndrome.
Phosphoserine acid phosphatase (PSPH) RNA | 2 years
  PSPH RNA level will be detected by fluorescence quantitative PCR in PDR group, SKYD group and NC group.
Phosphoserine acid phosphatase (PSPH) RNA in the cell models of disease-TCM syndrome | 2 years
  PSPH RNA level will be detected by fluorescence quantitative PCR in the cell models of disease-TCM syndrome.
Serine | 2 years
  Serine levels will be measured by targeted metabonomics in PDR group, SKYD group and NC group.
the differences of metabonomics in the cell models of disease-TCM syndrome | 2 years
  The differences of metabonomics in blood, urine and tongue coating will be detected by metabonomics in the cell models of disease-TCM syndrome.
the differences of transcriptomics in the cell models of disease-TCM syndrome | 2 years
  The differences of transcriptomics in blood, urine and tongue coating will be detected by transcriptomics in the cell models of disease-TCM syndrome.
the differences of metabonomics | 2 years
  The differences of metabonomics in blood, urine and tongue coating will be detected by metabonomics in PDR group, SKYD group and NC group.
the differences of proteomics in the cell models of disease-TCM syndrome | 2 years
  The differences of proteomics in blood, urine and tongue coating will be detected by proteomics in the cell models of disease-TCM syndrome.
the differences of transcriptomics | 2 years
  The differences of transcriptomics in blood, urine and tongue coating will be detected by transcriptomics in PDR group, SKYD group and NC group.
the differences of proteomics | 2 years
  The differences of proteomics in blood, urine and tongue coating will be detected by proteomics in PDR group, SKYD group and NC group.
Malondialdehyde (MDA) in the cell models of disease-TCM syndrome | 2 years
  Determination of MDA content by thiobarbituric acid method in the cell models of disease-TCM syndrome.
Malondialdehyde (MDA) | 2 years
  Determination of MDA content by thiobarbituric acid method in PDR group, SKYD group and NC group.
Superoxide Dismutase (SOD) in the cell models of disease-TCM syndrome. | 2 years
  Determination of SOD activity by xanthine oxidase method in the cell models of disease-TCM syndrome.
Superoxide Dismutase (SOD) | 2 years
  Determination of SOD activity by xanthine oxidase method in PDR group, SKYD group and NC group.
Peroxynitrite anion (ONOO-) in the cell models of disease-TCM syndrome | 2 years
  ONOO- will be detected by ELISA in the cell models of disease-TCM syndrome.
Peroxynitrite anion (ONOO-) | 2 years
  ONOO- will be detected by ELISA in PDR group, SKYD group and NC group.
Nicotinamide Adenine Dinucleotide Phosphate (NADPH) the cell models of disease-TCM syndrome | 2 years
  NADPH will be detected by ELISA in the cell models of disease-TCM syndrome.
Nicotinamide Adenine Dinucleotide Phosphate (NADPH) | 2 years
  NADPH will be detected by ELISA in PDR group, SKYD group and NC group.
Glutathione (GSH) in the cell models of disease-TCM syndrome. | 2 years
  GSH will be detected by ELISA in the cell models of disease-TCM syndrome.
Glutathione (GSH) | 2 years
  GSH will be detected by ELISA in PDR group, SKYD group and NC group.
3-phosphoglycerate dehydrogenase（PHGDH） in the cell models of disease-TCM syndrome | 2 years
  PHGDH will be detected by ELISA in the cell models of disease-TCM syndrome.
3-phosphoglycerate dehydrogenase（PHGDH） | 2 years
  PHGDH will be detected by ELISA in PDR group, SKYD group and NC group.
Threonine in the cell models of disease-TCM syndrome | 2 years
  Threonine levels will be measured by targeted metabonomics in the cell models of disease-TCM syndrome.
Threonine | 2 years
  Threonine levels will be measured by targeted metabonomics in PDR group, SKYD group and NC group.
Glycine in the cell models of disease-TCM syndrome | 2 years
  Glycine levels will be measured by targeted metabonomics in the cell models of disease-TCM syndrome.
Glycine | 2 years
  Glycine levels will be measured by targeted metabonomics in PDR group, SKYD group and NC group.
The clinical TCM scores of SKYD | 2 years
  The minimum value is 0 and maximum value is 35, and higher scores mean a worse outcome.
The clinical TCM scores of PDR | 2 years
  The minimum value is 0 and maximum value is 44, and higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Dongzhimen Hospital, Beijing, Dongcheng, China